CLINICAL TRIAL: NCT01208389
Title: A Follow-On Study to Evaluate the Safety of Re-Administration of Adeno-Associated Viral Vector Containing the Gene for Human RPE65 [AAV2-hRPE65v2] to the Contralateral Eye in Subjects With Leber Congenital Amaurosis (LCA) Previously Enrolled in a Phase 1 Study
Brief Title: Phase 1 Follow-on Study of AAV2-hRPE65v2 Vector in Subjects With Leber Congenital Amaurosis (LCA) 2
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Spark Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAV2-hRPE65v2-102; 10-007752 (Other: Children's Hospital of Philadelphia)
Record Dates: First submitted 2010-09-22; First posted 2010-09-24 (Estimated); Last update posted 2025-04-29 (Actual); Status verified 2024-12

CONDITIONS: Leber Congenital Amaurosis
MeSH Terms: conditions — Leber Congenital Amaurosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- voretigene neparvovec-rzyl (AAV2-hRPE65v2) (Experimental): Administration of study agent (AAV2-hRPE65v2) to the previously, uninjected contralateral eye:
  Interventions: Biological: voretigene neparvovec-rzyl

INTERVENTIONS:
Biological: voretigene neparvovec-rzyl — One time, subretinal administration of 1.5E11 vg AAV2-hRPE65v2 vector in 300 microliters to the contralateral, previously uninjected eye.
  Other Names: AAV2-hRPE65v2

SUMMARY:
The study is a follow-on to a Phase 1 dose-escalation and safety study.

DETAILED DESCRIPTION:
The study is a follow-on to a Phase 1 dose-escalation and safety study (closed to enrollment as of June 2009). Up to twelve adults and children with a molecular diagnosis of biallelic RPE65 mutations, who have participated in the earlier Phase 1 study, and who meet all study eligibility criteria, will receive AAV2-hRPE65v2 vector in the previously uninjected, contralateral eye to evaluate the safety of bilateral, sequential subretinal administration of AAV2-hRPE65v2.

ELIGIBILITY:
Inclusion Criteria:

* Prior participation in Phase 1 study with unilateral, subretinal administration of AAV2-hRPE65v2.
* Visual acuity equal to or greater than light perception.
* Sufficient viable retinal cells in contralateral, previously uninjected eye, as determined by non-invasive means, such as optical coherence tomography (OCT) and/or ophthalmoscopy. Must have either: 1) an area of retina within the posterior pole of > 100 µm shown on OCT; 2) ≥ 3 disc areas of retina without atrophy or pigmentary degeneration within the posterior pole; or 3) remaining visual field within 50 degrees of fixation.
* Willingness to adhere to protocol and long-term follow-up as evidenced by written informed consent or parental permission and subject assent (where applicable).

Exclusion Criteria:

* Unable or unwilling to meet requirements of the study.
* Participation in any other study of an investigational drug within the past six months.
* Use of retinoid compounds or precursors that could potentially interact with the biochemical activity of the RPE65 enzyme; individuals who discontinue use of these compounds for 18 months may become eligible.
* Prior intraocular surgery within six months.
* Known sensitivity to medications planned for use in the peri-operative period.
* Pre-existing eye conditions, such as glaucoma, or complicating systemic diseases that would preclude the planned surgery or could interfere with the interpretation of study. Complicating systemic diseases would include those in which the disease itself, or the treatment for the disease, can alter ocular function. Examples are malignancies whose treatment could affect central nervous system function (for example: radiation treatment of the orbit; leukemia with CNS/optic nerve involvement). Subjects with diabetes or sickle cell disease would be excluded if they had any manifestation of advanced retinopathy (e.g. macular edema or proliferative changes). Also excluded would be subjects with immunodeficiency (acquired or congenital) as there could be susceptibility to opportunistic infection (such as CMV retinitis).
* Individuals of childbearing potential who are pregnant or unwilling to use effective contraception for four months following vector administration.
* Any other condition that would not allow the potential subject to complete follow-up examinations during the course of the study and, in the opinion of the investigator, makes the potential subject unsuitable for the study.
* Subjects will NOT be excluded based on their gender, race, or ethnicity.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2010-11 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Adverse events as a measure of safety and tolerability | 15 years
  The primary outcome measures are safety and tolerability. Secondary outcome measure(s) include changes in visual function as measured by subjective, psychophysical tests and by objective, physiologic tests.

SECONDARY OUTCOMES:
Visual acuity | 15 years
  The primary outcome measures are safety and tolerability. Secondary outcome measure(s) include changes in visual function as measured by subjective, psychophysical tests and by objective, physiologic tests.
Visual field | 15 years
  The primary outcome measures are safety and tolerability. Secondary outcome measure(s) include changes in visual function as measured by subjective, psychophysical tests and by objective, physiologic tests.
Pupillary light response | 15 years
  The primary outcome measures are safety and tolerability. Secondary outcome measure(s) include changes in visual function as measured by subjective, psychophysical tests and by objective, physiologic tests.
Mobility testing | 15 years
  The primary outcome measures are safety and tolerability. Secondary outcome measure(s) include changes in visual function as measured by subjective, psychophysical tests and by objective, physiologic tests.
Full-field light threshold sensitivity testing | 15 years
  The primary outcome measures are safety and tolerability. Secondary outcome measure(s) include changes in visual function as measured by subjective, psychophysical tests and by objective, physiologic tests.
Contrast sensitivity | 15 years
  The primary outcome measures are safety and tolerability. Secondary outcome measure(s) include changes in visual function as measured by subjective, psychophysical tests and by objective, physiologic tests.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Director, Study Director — Spark Therapeutics, Inc.
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maguire AM, Simonelli F, Pierce EA, Pugh EN Jr, Mingozzi F, Bennicelli J, Banfi S, Marshall KA, Testa F, Surace EM, Rossi S, Lyubarsky A, Arruda VR, Konkle B, Stone E, Sun J, Jacobs J, Dell'Osso L, Hertle R, Ma JX, Redmond TM, Zhu X, Hauck B, Zelenaia O, Shindler KS, Maguire MG, Wright JF, Volpe NJ, McDonnell JW, Auricchio A, High KA, Bennett J. Safety and efficacy of gene transfer for Leber's congenital amaurosis. N Engl J Med. 2008 May 22;358(21):2240-8. doi: 10.1056/NEJMoa0802315. Epub 2008 Apr 27. PMID 18441370
- [Background] Maguire AM, High KA, Auricchio A, Wright JF, Pierce EA, Testa F, Mingozzi F, Bennicelli JL, Ying GS, Rossi S, Fulton A, Marshall KA, Banfi S, Chung DC, Morgan JI, Hauck B, Zelenaia O, Zhu X, Raffini L, Coppieters F, De Baere E, Shindler KS, Volpe NJ, Surace EM, Acerra C, Lyubarsky A, Redmond TM, Stone E, Sun J, McDonnell JW, Leroy BP, Simonelli F, Bennett J. Age-dependent effects of RPE65 gene therapy for Leber's congenital amaurosis: a phase 1 dose-escalation trial. Lancet. 2009 Nov 7;374(9701):1597-605. doi: 10.1016/S0140-6736(09)61836-5. Epub 2009 Oct 23. PMID 19854499
- [Background] Simonelli F, Maguire AM, Testa F, Pierce EA, Mingozzi F, Bennicelli JL, Rossi S, Marshall K, Banfi S, Surace EM, Sun J, Redmond TM, Zhu X, Shindler KS, Ying GS, Ziviello C, Acerra C, Wright JF, McDonnell JW, High KA, Bennett J, Auricchio A. Gene therapy for Leber's congenital amaurosis is safe and effective through 1.5 years after vector administration. Mol Ther. 2010 Mar;18(3):643-50. doi: 10.1038/mt.2009.277. Epub 2009 Dec 1. PMID 19953081
- [Background] Bennett J, Ashtari M, Wellman J, Marshall KA, Cyckowski LL, Chung DC, McCague S, Pierce EA, Chen Y, Bennicelli JL, Zhu X, Ying GS, Sun J, Wright JF, Auricchio A, Simonelli F, Shindler KS, Mingozzi F, High KA, Maguire AM. AAV2 gene therapy readministration in three adults with congenital blindness. Sci Transl Med. 2012 Feb 8;4(120):120ra15. doi: 10.1126/scitranslmed.3002865. PMID 22323828
- [Derived] Fischer MD, Simonelli F, Sahni J, Holz FG, Maier R, Fasser C, Suhner A, Stiehl DP, Chen B, Audo I, Leroy BP; PERCEIVE Study Group. Real-World Safety and Effectiveness of Voretigene Neparvovec: Results up to 2 Years from the Prospective, Registry-Based PERCEIVE Study. Biomolecules. 2024 Jan 17;14(1):122. doi: 10.3390/biom14010122. PMID 38254722
- [Derived] Bennett J, Wellman J, Marshall KA, McCague S, Ashtari M, DiStefano-Pappas J, Elci OU, Chung DC, Sun J, Wright JF, Cross DR, Aravand P, Cyckowski LL, Bennicelli JL, Mingozzi F, Auricchio A, Pierce EA, Ruggiero J, Leroy BP, Simonelli F, High KA, Maguire AM. Safety and durability of effect of contralateral-eye administration of AAV2 gene therapy in patients with childhood-onset blindness caused by RPE65 mutations: a follow-on phase 1 trial. Lancet. 2016 Aug 13;388(10045):661-72. doi: 10.1016/S0140-6736(16)30371-3. Epub 2016 Jun 30. PMID 27375040